CLINICAL TRIAL: NCT02893956
Title: Does Postural Support During Echocardiography Modify Hemodynamic Features and Discomfort Induced by the Examination in Very Premature Neonates?
Brief Title: Conditions of Realization of the Echocardiography in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 9252
Record Dates: First submitted 2016-07-21; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-08

CONDITIONS: Premature Newborn
Keywords: Echocardiography; postural support; preterm neonate
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- echocardiography with postural support then standard condition (Experimental): the first echocardiography (ultrasound) is performed with a postural support then the second echocardiography is performed with standard condition
  Interventions: Procedure: echocardiography with postural support; Procedure: echocardiography with standard condition (usual)
- echocardiography with standard condition then support postural (Active Comparator): the first echocardiography (ultrasounds) is performed with standard condition (usual) and the second echocardiography is performed with a postural support
  Interventions: Procedure: echocardiography with postural support; Procedure: echocardiography with standard condition (usual)

INTERVENTIONS:
Procedure: echocardiography with postural support
Procedure: echocardiography with standard condition (usual)

SUMMARY:
Experimental nociceptive stimulation of the fetus and neonate induces pulmonary artery vasoconstriction. The investigators assessed whether echocardiography for Ductus arteriosus screening may generate this hemodynamic response and whether postural support would be able to modulate it.

Study design

Prospective, single center, randomized study in less than 29 weeks of gestation neonates, with a post natal age < 48 hours, and requiring invasive mechanical ventilation.

Crossover design with order of echocardiographies determined by computer randomization: in one group ultrasounds are performed with postural support, than standard conditions, in the other, ultrasounds are performed in standard conditions than with postural support.

The objective of the study is to assess the ratio of the acceleration time/ejection time of pulmonary arterial flow.

The others objectives are to assess echocardiographic-Doppler features (ductus arteriosus shunt pattern, pulmonary flow pattern, estimated systolic pulmonary arterial pressure, right and left ventricular functions using tissue Doppler imaging and speckle-tracking echocardiography), pain assessment with a clinical scale and heart rate variability analysis.

ELIGIBILITY:
Inclusion Criteria:

* Newborn than 30 weeks of gestation neonates,
* Newborn with a post natal age < 48 hours,
* Newborn requiring invasive mechanical ventilation.
* Signed consent form of parent

Exclusion Criteria:

-

Ages: 1 Minute to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
value of the ratio of the acceleration time of pulmonary arterial flow. | up to 1 hour
  for each echocardiography (support condition and postural support)
value of the ejection time of pulmonary arterial flow | up to 1 hour
  for each echocardiography (support condition and postural support)

SECONDARY OUTCOMES:
pain assessment with a clinical scale | up to 1 hour
  assessment of the pain with a practical behavioral observation scale
number of participant with a Patent ductus arteriosus shunt | up to 2 hours
systolic pulmonary arterial pressure | up to 2 hour

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No